CLINICAL TRIAL: NCT02753556
Title: ScreenFlow: Strategy for Finding Cases of Moderate-to-Severe COPD
Status: Completed | Type: Observational
Sponsor: Dimagi Inc. (Industry)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HHSN268201400046C
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; ScreenFlow; Screening; Lung Disease; Mobile Health; Peak Flow Meter; Usability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ScreenFlow is a chronic obstructive pulmonary disease (COPD) screening tool currently being studied and iteratively developed that incorporates a questionnaire administered on a tablet and data from a digital peak flow meter to calculate a risk score to identify the risk of developing moderate-to-severe COPD for the participant. The purpose of this study is to assess the usability of ScreenFlow deployed as a free-standing kiosk and observe where users encounter trouble navigating the system. The kiosk will be situated in a public area of a hospital where passersby can approach and fill out a ScreenFlow survey if they meet the eligibility criteria. A subset of participants will be asked to participate in a follow-up questionnaire about their experience using the system and about any follow-up action they may have taken caused by their results from the ScreenFlow screening.

DETAILED DESCRIPTION:
This is a cross-sectional study to determine the usability of ScreenFlow deployed as a kiosk. As such, everyone who uses ScreenFlow will be asked to complete a brief questionnaire on its features including visual appeal and ease of use. Additionally, a subset of 36 subjects whose estimated ScreenFlow risk of moderate-to-severe COPD is high will be asked to participate in a follow up phone questionnaire to ascertain, a) whether screening results were discussed with the subjects' health provider, b) impact of the ScreenFlow results on health behavior, c) whether the individual shared the ScreenFlow result with his/her health provider (or intention to share the result), and d) any action that may have been taken by the medical provider after the provider received the report.

The ScreenFlow platform will be available in a common area of Boston Medical Center over the course of six weeks, under the supervision of a study staff member. The platform will be available to the public during regular business hours from Monday to Friday. Subjects will complete a ScreenFlow screening by answering some questions, watching a video and performing peak flow measurement as instructed in the video. They will be given a report of the ScreenFlow result indicating whether there is a high probability of having moderate to severe COPD. Over six weeks, approximately 3600 patients should come in contact with the kiosk. Conservatively, we estimate that if 10% of them use it, we will have 360 users, of which 10% may have a high risk score on screening. This will give the desired sample size of 36 patients for the phone based follow-up interview.

Thirty-six subjects will give their feedback through a phone based follow-up interview with a study staff member to assess how ScreenFlow may have influenced their subsequent medical care. We will consent 36 subjects for these follow-up calls, with the expectation that some may be difficult to reach or may decline to participate in the follow-up call.

In the interview we will ask whether the participants discussed COPD with their primary care providers, and the extent to which their care may have been influenced by this screening result. For those who have not had the opportunity to share results with their provider by the time of the follow-up call, we will ask about the effect of the positive screening result on their perception of COPD risk, intention to notify their provider, and health behavior.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older, able to use tablet

Exclusion Criteria:

* History of pneumothorax or collapsed lung, surgery in the past 6 months (oral, eye, chest, abdomen), non-English speaking, signs and symptoms of an active upper respiratory tract infection, legally blind and/or deaf

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from which possible participants will self-select is of people that pass through the pharmacy entrances at the Boston Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of positive ScreenFlow screens among participants that use system | Six weeks
  Out of the entirety of screening results for all participants that use the ScreenFlow system during the study, calculation of the proportion of "positive" screens

SECONDARY OUTCOMES:
Qualitative feedback on the usability of the ScreenFlow system | Six weeks
  Each participant that uses the ScreenFlow system will be asked to complete a qualitative survey upon completion of the ScreenFlow questionnaire. The survey will focus on the user experience and usability of the ScreenFlow system.
Click-based usability testing of the ScreenFlow interface | Six weeks
  During each session a participant completes using the ScreenFlow system, we will track each touch on the tablet screen, including the time it takes for a user to make each touch. This will provide input into questions that may be confusing to users, and interface designs that may not be intuitive.
Proportion of adults exposed to the ScreenFlow system that actually use it | Six weeks
  We will track the number of adults that are "exposed" wherein they pass by or see the ScreenFlow kiosk, and also keep track of how many "exposed" adult then opt to approach and use the system.

IPD SHARING:
Plan to Share IPD: No